CLINICAL TRIAL: NCT00557778
Title: Education and Awareness Program Targeting the Assessment of Adherence of the Treatment of Dyslipidemia
Acronym: PRECAVER
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Dr. Jose Eduardo Neves/Medical Director, AstraZeneca
Other Study IDs: NIS-CBR-CRE-2007/1
Record Dates: First submitted 2007-11-13; First posted 2007-11-14 (Estimated); Last update posted 2011-04-28 (Estimated); Status verified 2011-04

CONDITIONS: Patients With Dyslipidemia
Keywords: prevention; dyslipidemia
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Receives treatment with rosuvastatin, according to International and National Guidelines on hypercholesterolemia.
- Group 2: Receives the same treatment as group 1 and information on health improvement, diet and exercises applied to the disease that is being treated. The positive impact of the information upon treatment will be statistically evaluated.

SUMMARY:
Evaluate the benefit (rate of adherence to the treatment), based on the LDL-C reduction in the group that will be exposed to the program of reinforcement of orientation aimed to the patients, compared to the control group, both in previous use of rosuvastatin.

ELIGIBILITY:
Inclusion Criteria:

* Subjects eligible for the treatment of dyslipidemia with statins according the current guidelines NCEP ATPIII and IV Brazilian Guidelines of Dyslipidemia and Atherosclerosis Prevention.
* Patients with previous use of rosuvastatin for, at least, 15 days and, for no longer than12 months prior to the inclusion in the study.

Exclusion Criteria:

Pregnancy and childbearing

* History of severe hypersensitivity (including myopathy) to other HMG-CoA reductase inhibitors.
* Subjects with indication of use of cyclosporine and other associations of other lipid lowering drugs.
* Subjects with underlying diseases that may influence lipid levels (i.e. uncontrolled hypothyroidism defined as a Thyroid stimulating hormone (TSH) > 1.5 times upper level of normality (ULN) at Visit 1, AIDS, transplanted subjects, etc).
* History of drug and alcohol abuse.
* Current active liver disease or hepatic failure or elevations in ALT >3 times the ULN.
* Elevation of CPK > 3 times the ULN.
* Elevation in the seric creatinine > 2,0 mg / dL.
* History of malignancy in the last 5 years, except basal cell or squamous cell carcinoma of the skin (women with a history of Cervical dysplasia must be included, unless they have t3 clear consecutive Papanicolaou (Pap) smears , before the entry in the study).
* Any other known clinical condition that, in the opinion of the investigator, may compromise the subject's safety.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinic
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2007-11; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Assess the LDL-C reduction in the group exposed to the educational program compared to the group with routine orientation

SECONDARY OUTCOMES:
Assess cardiovascular risk through Framingham's score, · · Identify personal characteristics of the study population regarding their health, compile demographic characteristics regarding education, economic and cultural status.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Eduardo Neves, MD, Study Director — AstraZeneca Brazil Ltda; Francisco Jose Saraiva, MD, Principal Investigator — PUC-Campinas
Locations (1):
- Research Site, Campinas, São Paulo, Brazil